CLINICAL TRIAL: NCT07320963
Title: A Prospective, Single-Arm, Phase Ib/II Clinical Trial of Chidamide in Combination With Toripalimab and Anlotinib in Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma Who Have Failed at Least One Prior Line of Therapy
Brief Title: Chidamide in Combination With Toripalimab and Anlotinib in Recurrent/Metastatic Nasopharyngeal Carcinoma.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huiqiang Huang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-Q113
Record Dates: First submitted 2025-12-02; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: HDACi; PD-1 antibody; NPC; chidamide; anti-angiogenesis
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; toripalimab; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide , Toripalimab and Anlotinib (Experimental)
  Interventions: Drug: Chidamide; Biological: Toripalimab; Drug: Anlotinib

INTERVENTIONS:
Drug: Chidamide — Phase Ib: Dose selection based on study progression (15 mg, 20 mg, or 30 mg). Phase II: PR2D Timing: Orally 30 minutes after dinner, twice weekly (e.g., Days 1, 4, 8, 11, 15, 18 of each 3-week cycle), with ≥3 days between doses.
  Duration: Until disease progression or unacceptable toxicity, up to 24 months.
Biological: Toripalimab — Fixed Dose: 240 mg per infusion. Timing: Intravenous infusion over 30 minutes on Day 1 of each 3-week cycle. Duration: Until disease progression or unacceptable toxicity, up to 24 months.
Drug: Anlotinib — Timing: Orally once daily before breakfast, Days 1-14 of each 3-week cycle. Duration: Until disease progression or unacceptable toxicity, up to 24 months.

SUMMARY:
To explore and evaluate the dose-limiting toxicity (DLT) profile of the fixed-dose combination of toripalimab, anlotinib, and chidamide in patients with recurrent/metastatic nasopharyngeal carcinoma (R/M NPC), and to determine the maximum tolerated dose (MTD) of chidamide, thereby informing subsequent clinical dosing regimens.

To assess the objective response rate (ORR) of the combination regimen in this patient population.

ELIGIBILITY:
Inclusion Criteria:

- 1. Age: ≥18 years and ≤70 years, gender unrestricted. 2. Diagnosis: Histologically/pathologically confirmed metastatic nasopharyngeal carcinoma (NPC) that has failed at least one prior line of therapy (including cisplatin-containing regimens) or is intolerant to existing therapies (relapse within 6 months after completion of adjuvant/neoadjuvant concurrent chemoradiotherapy is eligible).

3. Performance Status: ECOG performance status 0-1. Measurable Disease: At least one measurable lesion per RECIST 1.1 criteria. 4. Prior Immunotherapy:

Patients who have received PD-1, PD-L1, PD-L2, or CTLA-4 inhibitors, or other therapies targeting T-cell co-stimulation/checkpoint pathways:

Must have achieved complete response (CR), partial response (PR), or stable disease (SD) ≥6 months during treatment.

Only one prior immunotherapy regimen is allowed (e.g., neoadjuvant and adjuvant regimens using the same immunotherapy are considered one regimen).

Switching to a different immunotherapy regimen for non-immunotherapy-related progression is permissible if cumulative SD duration ≥6 months.

6. Organ Function:

Hematology:

ANC ≥1.5×10⁹/L, PLT ≥75×10⁹/L, Hb ≥90 g/L. No blood product transfusion or growth factor support (e.g., G-CSF, EPO) within 2 weeks prior to screening.

Hepatology:

TBIL ≤1.5×ULN; ALT/AST ≤2.5×ULN (≤5×ULN if liver metastases present).

Renal Function:

Serum Cr ≤1.5×ULN or CrCl >60 mL/min.

Thyroid Function:

TSH, FT4, FT3 within CTC AE Grade 0-1. 7. Survival Expectancy: ≥3 months. 8. Informed Consent: Voluntary participation and signed written informed consent.

Exclusion Criteria:

1. Known severe hypersensitivity (≥Grade 3) to any monoclonal/polyclonal antibody, chidamide, or anlotinib components.
2. Necrotic lesions identified within 4 weeks prior to enrollment, with investigator-judged risk of major bleeding.
3. Chemotherapy, targeted therapy, or immunomodulatory agents (including thymosin, interferon, IL-2, etc.) within 2 weeks prior to enrollment.

   Washout period determined by clinical resolution of adverse events (AEs) and prior treatment regimens.
4. Palliative radiotherapy to localized lesions within 4 weeks prior to enrollment, unless the lesion is non-target and other measurable target lesions exist.
5. Grade ≥3 irAEs during prior immunotherapy.
6. Prior treatment with HDAC inhibitors or anti-angiogenic agents.
7. Urine protein ≥2+ or 24-hour urinary protein ≥1 g.
8. Systolic BP >140 mmHg or diastolic BP >90 mmHg despite treatment.
9. Persistent toxicity from prior antitumor therapy (per NCI CTCAE v5.0) >Grade 1, excluding: alopecia, Grade 2 fatigue, Grade 2 anemia, or asymptomatic lab abnormalities.
10. Symptomatic CNS metastases (e.g., edema, steroid requirement) or leptomeningeal disease.
11. Systemic immunosuppressive drugs (excluding topical/inhaled corticosteroids or physiological doses ≤10 mg/day prednisone equivalent) or corticosteroids for contrast allergy within 4 weeks prior to enrollment.
12. Active autoimmune diseases (e.g., interstitial pneumonia, colitis, thyroiditis) or history of severe autoimmune conditions requiring systemic therapy.

    Exceptions: Vitiligo, childhood asthma (resolved without treatment), or mild asthma managed without bronchodilators.
13. Ongoing anti-tuberculosis therapy or treatment within 1 year prior to screening.
14. Conditions requiring long-term immunosuppressive therapy or systemic corticosteroids at immunosuppressive doses.
15. Severe Cardiac Disease or Significant Cardiac Symptoms.
16. Other Circumstances Deemed Unsuitable by the Investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
MTD | 2 years
Objective Response Rate (ORR) | 2 years

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years
Duration of response (DoR) | 2 years
Overall Survival (OS) | 2 years

IPD SHARING:
Plan to Share IPD: No